CLINICAL TRIAL: NCT05103618
Title: Evaluating the Physiological and Psychological Effects of a Novel Meditation Technique on Cerebral Activity Measured With Functional Magnetic Resonance Imaging(fMRI) and F-18 Fluorodopa PET Imaging
Brief Title: Effect of Meditation and Controls and Subjects With Parkinson's Disease on Brain Activity Measured by fMRI With FDOPA
Acronym: FDOPAOM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: funding not obtained
Sponsor: Andrew Newberg (Other)
Responsible Party: Sponsor-Investigator, Andrew Newberg, Professor, Department of Integrative Medicine and Nutritional Sciences; Professor, Department of Radiology, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 21D.632
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease
Keywords: Alternative Medicine; Complementary Medicine; Parkinson's disease; Neurodegenerative Diseases; Idiopathic Parkinson's disease; Central Nervous System Diseases; Movement Disorders; [F-18] Fluorodopa; Magnetic Resonance Spectroscopy PET; Positron Emission Tomography; Dopaminergic Function
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Central Nervous System Diseases; Movement Disorders

STUDY DESIGN:
Intervention Model Description: This is an Open Label study. Subjects will be assigned a study number that will be used on the research files. Two group of couple pairs will be enrolled into this study: one group will be healthy couple pairs in which neither member has PD. The other couple pairs will include a female member with PD. For subjects who are enrolled in the meditation training programs couple pairs in which the female member has PD may be assigned to an active group or a waitlist control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Healthy Control Couple Pairs (Active Comparator): All healthy control subjects, 6 couple pairs (12 subjects) healthy controls in which neither member has Parkinson's Disease will receive a baseline and follow up FDOPA PET scan. All subjects will be asked to complete the surveys. The control group will receive training materials in the practice of OM which the couple will be asked to practice for the next 2-3 months. The couple-pair will begin the OM practice initially (in between the baseline and follow up scans. FDOPA scans and surveys will be conducted with both members of the couple pair at approximately 2-3 months.
  Interventions: Behavioral: OM Meditation
- Active Couple Pairs Parkinson's Group (Active Comparator): 15 Couple pairs (30 subjects) in which one female member has a diagnosis of PD.
  The female subject will undergo the baseline scan. Both members of the couple will complete surveys. The active group will receive training materials in the practice of OM which they will be asked to practice for the next 2-3 months The active couple-pair will begin the OM practice initially (in between the baseline and follow up). FDOPA scans will be conducted with female members with PD the couple pair at approximately 2-3 months.
  Interventions: Drug: [F-18] Fluorodopa Positron Emission Tomography; Behavioral: OM Meditation
- Waitlist Couple Pairs Parkinson's Group (Other): 15 Couple pairs (30 subjects) in which one female member has a diagnosis of PD. The female subject will undergo the baseline scan. Both members of the couple will complete surveys The waitlist period in which the female member with PD will continue to receive standard of care for those 2-3 months; who then receive follow up scan. After the follow up scan, the waitlist group may be trained in the practice of OM for the next two months (but there will not be an additional FDOPA scan). Couple-pairs in the waitlist group will be asked to complete surveys at baseline and follow up scan and again after completing the OM Meditation practice. Couple pairs will engage in OM Meditation together approximately 3-4 times a week after the baseline and follow up scans for 2-3 months but female subjects with PD will not receive and additional post OM Meditation FDOPA scan
  Interventions: Drug: [F-18] Fluorodopa Positron Emission Tomography

INTERVENTIONS:
Drug: [F-18] Fluorodopa Positron Emission Tomography — Subjects will receive FDOPA imaging at baseline and 2-3 months after practicing the OM Meditation for evaluation of the dopamine function, [F-18] Fluorodopa (FDOPA), dose (5-10 mCi, ± 20%) will be injected intravenously into an antecubital vein. In accordance with the standard imaging protocol for FDOPA; subjects will be pre-medicated with 200 mg of carbidopa orally approximately one hour prior to injection.
  Other Names: FDOPA PET/MRI
  Arms: Active Couple Pairs Parkinson's Group; Waitlist Couple Pairs Parkinson's Group
Behavioral: OM Meditation — Couple pairs will engage in OM Meditation together approximately 3-4 times a week approximately 2-3 months.
  Arms: Active Couple Pairs Parkinson's Group; Healthy Control Couple Pairs

SUMMARY:
The purpose of this research is to use 18 F Fluorodopa positron emission tomography (FDOPA PET) to measure dopamine function, and utilize magnetic resonance imaging (MRI) to measure inflammatory and oxidative stress markers in persons with Parkinson's disease.

The overall goal of this study will be to further the understanding of the effects of a novel meditation technique called orgasmic meditation (OM) on these neurophysiological parameters.

DETAILED DESCRIPTION:
The overall goal of this study is to further the understanding of the physiological and psychological effects and dopaminergic function of OM in couple pairs in a control group and in couples in which one member has Parkinson's disease (PD). This study will utilize F-18 Fluorodopa (FDOPA) positron emission tomography (PET) imaging which utilizes an experimental radioactive tracer called FDOPA which helps to evaluate the activity in the dopamine neurons in the brain. A secondary goal of this study is to determine whether undergoing OM meditation alters body or brain physiology, and to measure whether there is an effect on intimacy and sexual dysfunction in women with PD.

This study is designed to understand the changes that occurs when subjects undergo intense meditation or meditation induced by sensory stimulation and structured touch. This study is designed to allow researchers to understand the changes in couple-pairs that occur when subjects undergo a shared meditation practice. Since meditation practices are widely used by individuals, the Investigators hope that a better understanding of the effects of meditation practices will provide information regarding potential clinical uses.

80 subjects will be enrolled (6 healthy couple pairs) and 30 couple pairs in which one female member has PD. The Investigators will also for a 10% attrition to enroll a total of 72 subjects.

For evaluation of the dopamine function, [F-18] Fluorodopa (FDOPA), dose (5-10 millicurie (mCi), ± 20%) will be injected intravenously into an antecubital vein. Subjects will be premedicated with 200 mg of carbidopa orally approximately one hour prior to injection.

FDOPA has been available for over 30 years but has not been previously approved for commercial use by the FDA. The Investigators will be obtaining the FDOPA from the University of Pennsylvania cyclotron that has produced FDOPA for many Investigational New Drug applications (INDs) It will also be beneficial to assess whether there are specific changes in levels of different molecules that are related to energy consumption and oxidative stress. Proton MR spectroscopy (1H-MRS) has been previously performed in Parkinson's disease (PD) and parkinsonian syndromes to evaluate in vivo concentrations of basal ganglia and cerebral cortex metabolites such as N-acetylaspartate (NAA), choline (Cho), and creatine (Cr).

ELIGIBILITY:
Inclusion Criteria:(Control Group: 6 healthy, normal couple pairs)

1. No clinical diagnosis of PD
2. Age 25 years old and older
3. Physically independent, ambulatory
4. Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the period of pilot study. In addition, male subjects who have a partner of childbearing age should practice effective contraception.

Inclusion Criteria for Female Partner in Couple Pairs in Parkinson's Group who has Parkinson's Disease

1. Clinical diagnosis of PD in female partner
2. Age 30 years old and older
3. Physically independent, ambulatory
4. Hoehn and Yahr score of I-III inclusive.
5. On stable antiparkinsonian medication for at least one month
6. Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the period of pilot study. In addition, male subjects who have a partner of childbearing age should practice effective contraception.

Inclusion Criteria for Second Partner with No PD in Couple Pairs in Parkinson's Group

1. No clinical diagnosis of PD
2. Age 25 years old and older
3. Physically independent, ambulatory
4. Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the period of pilot study. In addition, male subjects who have a partner of childbearing age should practice effective contraception.

Exclusion Criteria: (In Control Couple Pairs and in Couple Pairs Group in which the Female member has PD)

1. Previous brain surgery.
2. Cognitive impairment by evaluation or known score on Mini-Mental Status examination of 25 or lower.
3. Wheelchair-bound or bed-ridden, non-ambulatory.
4. Intracranial abnormalities that may complicate interpretation of the brain scans (e.g., stroke, tumor, vascular abnormality affecting the target area).
5. Diagnosis of traumatic brain injury with significant impairment.
6. Any medical disorder or physical condition that could reasonably be expected to interfere with the assessment of parkinsonian syndrome symptoms, or with any of the study assessments including the PET-MRI imaging.
7. No metal in their body that would prevent MRI scanning (as determined by the PI).
8. Subjects with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate.
9. Subjects with current alcohol or drug abuse.
10. Pregnant or lactating women.
11. Enrollment in active clinical trial/ experimental therapy within the prior 30 days.
12. Pending surgery during the course of the study.
13. History of thrombocytopenia or clotting disorders.
14. Cancer patients receiving active chemotherapy.
15. History of uncontrolled diabetes and/or thyroid conditions.
16. History of severe kidney disease (if a subject reports this problem, a serum creatinine will be checked to assess glomerular filtration rate (GFR) and if it is less than 30, they will be excluded).

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07-08 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-07-21 (Actual)

PRIMARY OUTCOMES:
FDOPA PET | Subjects will receive FDOPA imaging at baseline
  The primary outcome measure will be the specific uptake values at 3 to 4 hours post administration, when the distribution of FDOPA has approached a transient, near equilibrium like state that reflects the ratio of k3/k4, which is related to binding potential. This allows for a quantitative assessment of dopamine activity.
FDOPA PET | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes in Dopaminergic Function.]
  The primary outcome measure will be the specific uptake values at 3 to 4 hours post administration, when the distribution of FDOPA has approached a transient, near equilibrium like state that reflects the ratio of k3/k4, which is related to binding potential. This allows for a quantitative assessment of dopamine activity.

OTHER OUTCOMES:
The Speilberger State Trait Anxiety Inventory | These will be obtained initially at baseline or the first imaging appointment
  The Spielberger State Trait Anxiety Inventory (STAI-Y) Contains a total of 40 questions, The range of possible scores for the STAI-Y form varies from a minimum score of 20 to a maximum score of 80 on both the STAI-Trait and STAI-State subscales. STAI scores are commonly classified as no or low anxiety score range (20-37), moderate anxiety score range (38-44), and high anxiety score range of (45-80). A higher score indicates more anxiety.half of which relate to the way subjects are feeling at the moment and half of which ask them to describe how they usually feel.
The Speilberger State Trait Anxiety Inventory | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes
  The Spielberger State Trait Anxiety Inventory (STAI-Y) Contains a total of 40 questions, The range of possible scores for the STAI-Y form varies from a minimum score of 20 to a maximum score of 80 on both the STAI-Trait and STAI-State subscales. STAI scores are commonly classified as no or low anxiety score range (20-37), moderate anxiety score range (38-44), and high anxiety score range of (45-80). A higher score indicates more anxiety.half of which relate to the way subjects are feeling at the moment and half of which ask them to describe how they usually feel.
The Profile of Moods Scale | These will be obtained initially at baseline or the first imaging appointment
  Profile of Mood States is a standardized self-report inventory will be administered to evaluate changes in mood, current state or traits. is a psychological rating scale used to assess transient, distinct mood states. The questionnaire contains 65 words that are rated on a scale of zero for not at all to 4 for extremely. There are 5 mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. A higher score for the total mood indicates a greater degree of mood disturbance.A Total Mood Disturbance (TMD) can be calculated by adding the raw scores from tension, depression, anger, fatigue and confusion and then subtracting the vigour score. This will give a value between -24 and 177, with lower scores indicative of people with more stable mood profiles.
The Profile of Moods Scale | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes
  Profile of Mood States is a standardized self-report inventory will be administered to evaluate changes in mood, current state or traits. is a psychological rating scale used to assess transient, distinct mood states. The questionnaire contains 65 words that are rated on a scale of zero for not at all to 4 for extremely. There are 5 mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. A higher score for the total mood indicates a greater degree of mood disturbance.A Total Mood Disturbance (TMD) can be calculated by adding the raw scores from tension, depression, anger, fatigue and confusion and then subtracting the vigour score. This will give a value between -24 and 177, with lower scores indicative of people with more stable mood profiles.
The Beck Depression Inventory | Subjects will be obtained initially at baseline or the first imaging appointment
  Beck Depression Inventory (Beck 1972) is a 21 question self report inventory to access depression and changes in mood. The highest possible total for the whole test would be 63; the lowest possible score for the test would be zero. A higher score indicates worse symptoms of depression and mood.
The Beck Depression Inventory | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes
  Beck Depression Inventory Beck 1972) is a 21 question self report inventory to access depression and changes in mood. The highest possible total for the whole test would be 63; the lowest possible score for the test would be zero. A higher score indicates worse symptoms of depression and mood.
Marital Intimacy Questionnaire | Subjects will be obtained initially at baseline or the first imaging appointment
  The Marital Intimacy Questionnaire (MIQ) is a theory-based self-report questionnaire assessing 5 components of marital intimacy. Construct validity was established by examining the correlations of the MIQ with measures of marital satisfaction, perceived global intimacy, and communication intimacy, and discriminant validity by showing its ability to discriminate between maritally distressed and non-distressed couples. The MIQ is a 56-item, Likert-type questionnaire designed to measure communication styles and levels of intimacy among married or cohabitating couples.Subscales on communication, intimacy and satisfaction are correlated in couple-pairs.
Marital Intimacy Questionnaire | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes
  The Marital Intimacy Questionnaire (MIQ) is a theory-based self-report questionnaire assessing 5 components of marital intimacy. Construct validity was established by examining the correlations of the MIQ with measures of marital satisfaction, perceived global intimacy, and communication intimacy, and discriminant validity by showing its ability to discriminate between maritally distressed and non-distressed couples. The MIQ is a 56-item, Likert-type questionnaire designed to measure communication styles and levels of intimacy among married or cohabitating couples. Subscales on communication, intimacy and satisfaction are correlated in couple-pairs.
The Female Sexual Function Index | Subjects will be obtained initially at baseline or the first imaging appointment
  The Female Sexual Function Index (FSFI) is a 19-item questionnaire, has been developed as a brief, multidimensional self report instrument for assessing the key dimensions of sexual function in women. The Questionnaire described was designed and validated for assessment of female sexual function and quality of life in clinical trials or epidemiological studies.The Female Sexual Function Scale total score is the sum of the 6 domain/subscale scores and has a maximum score of 36. Higher scores indicate better functioning. A total score 26.0 has been validated as a cutoff score for diagnosing Female Sexual Dysfunction.
The Female Sexual Function Index | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes
  The Female Sexual Function Index (FSFI) is a 19-item questionnaire, has been developed as a brief, multidimensional self report instrument for assessing the key dimensions of sexual function in women. The Questionnaire described was designed and validated for assessment of female sexual function and quality of life in clinical trials or epidemiological studies.The Female Sexual Function Scale total score is the sum of the 6 domain/subscale scores and has a maximum score of 36. Higher scores indicate better functioning. A total score 26.0 has been validated as a cutoff score for diagnosing Female Sexual Dysfunction.
Parkinson's Disease Questionnaire-39 | Subjects will be obtained initially at baseline or the first imaging appointment
  Parkinson's Disease Questionnaire-39 (PDQ).is a self report inventory that will be used to access changes in Parkinson's Disease symptoms. The total score for the PDQ is the sum of the scores for the 20 items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero. Individual subscale scores for attention/concentration, retrospective memory, prospective memory, and planning/organization can also be generated by calculating the sum of specific sets of items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero.
Parkinson's Disease Questionnaire-39 | Change from Baseline at 60-90 days ( approximately 2-3 months) to access changes
  Parkinson's Disease Questionnaire-39 (PDQ).is a self report inventory that will be used to access changes in Parkinson's Disease symptoms. The total score for the PDQ is the sum of the scores for the 20 items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero. Individual subscale scores for attention/concentration, retrospective memory, prospective memory, and planning/organization can also be generated by calculating the sum of specific sets of items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD,MBA, Study Chair — TJU, Integrative Medicine and Nutritional Sciences
Locations (1):
- Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After each participant completes the study, study scan data will be shared with co-investigators; participants may receive a copy of each scan after study completion.
Supporting Information: CSR
Time Frame: Study scan report will be offered to the subject after subject completes study
Access Criteria: Access only to authorized research staff and study participants

DOCUMENTS (1):
  • Informed Consent Form (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/18/NCT05103618/ICF_001.pdf